CLINICAL TRIAL: NCT06600698
Title: Evaluate Safety and Efficacy of Daily Oral Angelica Gigas Nakai (AGN)-INM176 in Prostate Patients With Rising Plasma PSA (Phase I/II Trial)
Brief Title: Safety and Efficacy of AGN-INM176 in Prostate Patients With Rising PSA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Junxuan Lu, Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-24-010
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Angelica gigas Nakai; INM 176; Pharmacokinetics; Decursin; decursinol; prostate specific antigen (PSA)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a one-arm, sequential Phase I/II study to evaluate INM176. Phase I uses a 3+3 dose escalation design to find the recommended Phase 2 dose (RP2D) based on dose-limiting toxicities. Phase II includes two stages: Stage 1 involves 13 subjects to test early efficacy; if ≥1 responds (PSA decline/stabilization), the study moves to Stage 2. Stage 2 enrolls 14 more subjects (total 27) to assess efficacy. A PSA response rate >5% is declared if ≥4 subjects show response. Safety and efficacy will be evaluated with descriptive statistics, linear mixed-effects models, and regression analyses for PK and biomarkers.
  Intervention Type: Drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INM176 Dose Escalation and Tolerability Assessment in phase I and efficacy assessment in phase II (Experimental): Phase I evaluates the safety and tolerability of INM176 using a dose escalation design. Participants will receive INM176 at the following dose levels: Dose Level -1 (400 mg/day), Dose Level 0 (800 mg/day), Dose Level +1 (1200 mg/day), and Dose Level +2 (1600 mg/day). The trial starts with 3 subjects at Dose Level 0. If none experience dose-limiting toxicity (DLT), 3 more subjects will be escalated to Dose Level +1. If one subject at Dose Level 0 experiences DLT, 3 additional subjects will be enrolled at the same level. Dose Level -1 is considered the maximum tolerated dose if 2 or more of 6 subjects experience DLT at Dose Level 0. The recommended Phase II dose (RP2D) may be the MTD or Dose Level +2 if no DLT is observed.
  Phase II measures changes in Prostate-Specific Antigen (PSA) levels from baseline to after 6 cycles of treatment at the Recommended Phase II Dose (RP2D). PSA level declines from baseline or stays same will be recorded as a positive responder to INM176.
  Interventions: Drug: INM176

INTERVENTIONS:
Drug: INM176 — The active ingredient INM176 was prepared using a proprietary technology to extract AGN with ethanol and powderize with cellulose into a finished granular powder product that is 1/5 the weight of the raw herbal root. This product was chosen because its close match with the AGN extracts studied in the TRAMP model in the phytochemical profiles. It will be donated from the manufacturer Nutragen Co., Ltd. Korea.

SUMMARY:
This Phase I/II open-label trial aims to evaluate the safety and efficacy of the herbal supplement INM176 in patients with a history of prostate cancer or low-risk disease under active surveillance. The study will determine the recommended Phase II dose (RP2D) and assess the efficacy of INM176 in stabilizing or decreasing plasma PSA levels in post-radical prostatectomy (RP) and post-radiation therapy (RT) patients with rising PSA levels.

DETAILED DESCRIPTION:
The study is designed as a Phase I/II open-label trial to assess the safety and preliminary efficacy of the herbal supplement INM176 in intercepting prostate cancer-specific PSA levels. The primary objective of the Phase I stage is to determine the recommended Phase II dose (RP2D) through a 3+3 dose escalation design while evaluating the safety of INM176 during a 4-week cycle for dose-limiting toxicities (DLTs) in patients with a history of prostate cancer or those under active surveillance for low-risk disease.

In the Phase II stage, the primary objective is to evaluate the efficacy of INM176 at the RP2D in stabilizing or reducing plasma PSA levels after six cycles of treatment in post-RP and post-RT patients experiencing a rise in PSA.

Secondary objectives include pharmacokinetic (PK) evaluations following the first dose (Cycle 1 Day 1) in both Phase I and Phase II subjects, with an additional PK assessment on Cycle 1 Day 28 for Phase I subjects and on Cycle 2 Day 1 for Phase II subjects. Acute and chronic exposure PK parameters (including Cmax and AUC) will be correlated with safety outcomes and prostate-specific antigen (PSA) efficacy measures, when applicable, stratified by CYP2C19 and CYP3A4 metabolizer status.

Additional secondary objectives include evaluation of PSA change from baseline at protocol-specified timepoints; immunophenotyping of blood natural killer (NK) cells and other immune cell subsets; assessment of NK functional activity, plasma IL-8, and select cytokines; and measurement of male hormones and hormone-binding proteins. These pharmacodynamic biomarkers will be analyzed in relation to PSA response and PK metrics, with assessments conducted according to Phase I and Phase II study schedules.

ELIGIBILITY:
Inclusion Criteria:

Phase I Inclusion Criteria

* Willingness and ability to give informed consent.
* Agree to comply with all study procedures and attend all study visits.
* Male aged >=40 years.
* History of prostate cancer diagnosis: Subjects with treated prostate cancer are eligible. Prior prostate cancer treatments must be clearly defined. Acceptable treatment modalities include surgery, radiation therapy, and previous use of antiandrogen therapy. Subjects with localized prostate cancer in low-risk group who were not on treatment or declined any treatment are eligible. Subjects with localized prostate cancer in the favorable intermediate-risk group who declined any treatment are eligible.
* Subjects must not be undergoing concurrent radiation therapy or androgen deprivation therapy (ADT) at the time of enrollment.
* ECOG performance status 0-2.
* Subjects must have normal liver and kidney function at baseline: Total bilirubin within normal institutional limits. AST(SGOT)/ALT(SGPT) < 2.5 X upper limit of normal (ULN). Creatinine < 1.5 ULN or creatinine clearance > 50 mL/min/1.73 m2. Adequate bone marrow function: Hgb ≥ 9.0 g/dL, Platelets ≥ 100 x 109/L, absolute neutrophil count of ≥ 1.0 x 109/L).International Normalized Ratio (INR), Prothrombin Time (PT), and Partial Thromboplastin Time (PTT)within normal institutional limits.
* Subjects and their partners must agree to use two medically accepted methods of contraception and must agree to continue use these methods during the trial and for at least one week after the last dose of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) withdrawal, spermicides only, or lactational amenorrhea are not acceptable methods of contraception.
* Subjects taking strong inhibitors or inducers of CYP3A4 or CYP2C19 must be evaluated for potential drug interactions with the study drug. Essential medications, such as statins, that cannot be discontinued may be allowed at the investigator's discretion.
* Subjects currently taking herbal supplements containing AGN extract, such as Cogni.Q, Decursinol-50, Ache Action, Fast-Acting Joint Formula, must discontinue these or any other supplements containing these products at least 4 weeks prior to starting study drug.

Phase II Inclusion Criteria

* Willingness and ability to give informed consent.
* Agree to comply with all study procedures and attend all study visits.
* Male aged >=40 years.
* Histologically confirmed adenocarcinoma of prostate (neuroendocrine or small cell prostate cancer excluded).
* Any T stage, N0-1, M0, any Gleason grade.
* Subjects must meet one of the following: Post-radical prostatectomy (RP) and/or post-radiation therapy (RT), including those with local recurrence declining further treatment. Localized prostate cancer who declined any treatment after physician discussion.
* No distant metastases disease confirmed by imaging (CT or MRI and bone scan or prostate-specific PET scan such as PSMA PET scan or Axumin PET scan) within 5 years prior to enrollment.
* Blood PSA level rising over 2 consecutive tests within the past 6 months, at least one week apart, with values ≥ 0.1 ng/mL.
* Not currently receiving concurrent androgen deprivation therapy, and testosterone levels should be within a non-castrate range (>50 ng/dL).
* ECOG performance status 0-2.
* Subjects must have normal liver, kidney, and bone marrow function at baseline: Total bilirubin within institutional limits. AST(SGOT)/ALT(SGPT) < 2.5 X upper limit of normal (ULN). Creatinine < 1.5 ULN or creatinine clearance > 50 mL/min/1.73 m2. Adequate bone marrow function: Hgb ≥ 9.0 g/dL, Platelets ≥ 100 x 109/L, absolute neutrophil count ≥ 1.0 x 109/L.
* No evidence of any active secondary malignancy requiring ongoing treatment.
* Subjects must agree to use two medically accepted method of contraception and must agree to continue use this method while on the trial and through at least one week after the last dose of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) withdrawal, spermicides only, or lactational amenorrhea are not acceptable methods of contraception.
* Subjects taking strong inhibitors or inducers of CYP3A4 or CYP2C19 will be evaluated for potential drug interactions with the study drug. Essential medications, such as statins, that cannot be discontinued may be allowed at the investigator's discretion.
* Subjects currently taking herbal supplements containing AGN extract, including Cogni.Q, Decursinol-50, Ache Action, Fast-Acting Joint Formula, must discontinue these or any other supplements containing these products at least 4 weeks prior to starting study drug.
* Prior Phase I subjects: must have completed ≥90 days washout from the last investigational product dose and meet all of the following: no study-drug related AEs > Grade 1, hepatic and renal function tests within protocol-defined limits, and investigator confirmation of clinical stability.

Phase I and II Exclusion Criteria:

* Subjects with distant metastatic cancer. Node-positive prostate cancer patients are allowed after completion of treatment.
* Subjects who are receiving systemic treatments such as chemotherapy, androgen deprivation therapy (ADT) or anti-androgen therapy including LHRH agonist, antagonist, GNRH analogs, and antiandrogens, or immunotherapy (checkpoint inhibitor) or investigational agents.
* Participants will be excluded if they have any uncontrolled intercurrent illness at the discretion of the treating investigator. This may include, but is not limited to, the following conditions: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes mellitus (DM) with an HbA1C >9, uncontrolled asthma, or significant psychiatric illness that would limit compliance with study requirements.
* History of New York Heart Association Class III or IV heart failure, history of a myocardial infarction within 6 months, or any other cardiac-related problem that would be considered a contraindication for participation in the opinion of the treating physician.
* Any active secondary malignancy requiring treatment.
* Chronic kidney disease with calculated GFR <30 mL/min/1.73 m(2) using Cockcroft-Gault formula, or measured GFR <30 mL/min/1.73 m(2) using a 24-hour urine collection. The hospital's lab measured GFR can be used if a 24-hour collection is not possible.
* Subjects who are taking Warfarin/coumadin.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 45 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety of INM176 after 1, 2, 3,4, 5, and 6 cycles of exposure at RP2D | 10 months
  Safety will be assessed as the combined incidence of adverse events, abnormal safety blood tests, and abnormal ECG readings, expressed as the proportion of participants showing any of these safety concerns following 1, 2, 3, 4, 5, and 6 treatment cycles.
Efficacy of INM176 by Measuring PSA Level Changes After 6 Cycles of Treatment at the Recommended Phase II Dose (RP2D) | 10 months
  This outcome will assess the efficacy of INM176 by measuring changes in Prostate-Specific Antigen (PSA) levels from baseline to after 6 cycles of treatment at the Recommended Phase II Dose (RP2D). PSA levels will be monitored at baseline and following each treatment cycle, with a primary focus on the change observed after 6 cycles. The degree of PSA reduction will serve as an indicator of INM176's effectiveness in controlling or reducing prostate cancer activity.
Maximum Tolerated Dose (MTD) | 28 days
  The Maximum Tolerated Dose (MTD) is defined as the highest dose at which ≤1 of 6 participants experiences a dose-limiting toxicity (DLT) during Cycle 1 (28 days). Dose-limiting toxicities will be assessed according to CTCAE version 5.0.
Recommended Phase II Dose (RP2D) | 28 days
  The Recommended Phase II Dose (RP2D) will be determined based on overall safety and tolerability, observed dose-limiting toxicities, following dose escalation using a standard 3+3 design.
Dose-Limiting Toxicities (DLTs) | 28 days
  Dose-Limiting Toxicities (DLTs) are defined as adverse events or laboratory abnormalities that are considered to be related to the study treatment and occur during the first treatment cycle (28 days). DLTs will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The occurrence of DLTs will guide dose escalation decisions and help identify the Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D).

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States